CLINICAL TRIAL: NCT00106236
Title: Sapporo Fitness Club Trial (SFCT): A Randomized Controlled Trial to Test the Efficacy of Exercise at a Fitness Club for the Reduction of Cardiovascular Risk Factors
Brief Title: Efficacy of Exercise at a Fitness Club for Cardiovascular Risk Reduction
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sapporo Health Promotion Foundation (Other)
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: SHPCR-2003-1
Record Dates: First submitted 2005-03-21; First posted 2005-03-22 (Estimated); Last update posted 2009-07-14 (Estimated); Status verified 2005-03

CONDITIONS: Diabetes Mellitus; Hypertension; Hyperlipidemia
Keywords: Exercise; Fitness Club; Randomized Controlled Trial; Cardiovascular Risk Factor; Overweight; Inactivity
MeSH Terms: conditions — Diabetes Mellitus; Hypertension; Hyperlipidemias; Motor Activity; Overweight; Sedentary Behavior | interventions — Exercise

INTERVENTIONS:
Behavioral: exercise

SUMMARY:
The purpose of the study is to determine whether exercise has further beneficial effects on improving cardiovascular risk factors such as hypertension, high cholesterol level or diabetes mellitus, when added to the standard program of health check followed by life style recommendations.

DETAILED DESCRIPTION:
Multiple risk factors contribute to the causation of atherosclerotic cardiovascular disease. Past studies indicate that exercise exerts its protective effects on the disease through actions on multiple cardiovascular risk factors simultaneously; however, the studies focused on the effect of exercise predominantly on subjects with a single risk factor. Does exercise differentially act on various risk factors in the same subject? Do subjects with multiple risk factors respond differently to exercise than those predominantly with a single risk factor do? To our knowledge, this is the first large-scale study to test the efficacy of exercise on subjects with multiple risk factors. Exercise in fitness clubs has uniquely fitting features for middle to older aged people with multiple risk factors: access is relatively easy because there are usually many clubs throughout the city; the control of exercise intensity or heart rate is made precise, rendering exercise safer when treadmills or bicycles are used as a mainstay of aerobic exercise as in this study; and cardiac arrest, the most feared complication of exercise, will be most likely to be properly handled since in recent years the installment of automated external defibrillators has been increasingly popular in many clubs.

Comparison: Exercise vs. standard care comparison is to be made only for the first 6-month period. The second 6-month period is for follow-up and other purposes.

ELIGIBILITY:
Inclusion Criteria:

Body mass index (BMI) of 24.2-34.9 with 2 or more of the following risk factors:

* Resting systolic blood pressure of 130-179 mmHg
* Fasting blood glucose of 110-139 mg/dl, or HbA1c ≥ 5.8 when casual blood sugar is 140-199 mg/dl
* LDL-cholesterol of 120-219 mg/dl

Exclusion Criteria:

* Diastolic blood pressure of 110 mmHg or greater
* History of clinical heart disease or stroke
* Orthopedic problems that might interfere with exercise
* Dementia
* Abnormal exercise EKG test results
* Private physician's disapproval

Ages: 45 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 561
Dates: Start 2003-04; Study Completion 2004-04

PRIMARY OUTCOMES:
Systolic blood pressure
low-density lipoprotein cholesterol
hemoglobin A1c

SECONDARY OUTCOMES:
Body weight
waist circumference
diastolic blood pressure
HDL-cholesterol
triglyceride
casual blood glucose
high-sensitivity C-reactive protein
white blood cell count
estimated VO2max
bicycle time
leg muscle strength
health-related QOL (Quality of Life)

CONTACTS AND LOCATIONS:
Locations (1):
- Sapporo Health Promotion Center, Sapporo, Hokkaido, Japan

REFERENCES:
- [Background] Igarashi K, Fujita K, Yamase T, Morita N, Okita K, Satake K, Kanazawa N, Nishijima H. Sapporo Fitness Club Trial (SFCT)--design, recruitment and implementation of a randomized controlled trial to test the efficacy of exercise at a fitness club for the reduction of cardiovascular risk factor--. Circ J. 2004 Dec;68(12):1199-204. doi: 10.1253/circj.68.1199. PMID 15564707